CLINICAL TRIAL: NCT02301052
Title: Double Blind Randomized Placebo-control Trial of Allium Ampeloprasum Spp.Iranicum Cream Effect for the Management of Hemorrhoids Symptoms
Brief Title: Evaluation of Allium Ampeloprasum Spp.Iranicum Cream Effect for the Management of Hemorrhoids Symptoms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leyla Ghahramani, Shiraz university of medical sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-9377-7127
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids; Allium Ampeloprasum; herbal medicine; traditional persian medicine
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): placebo topical cream 2 cc twice daily for 3 weeks
  Interventions: Drug: placebo topical cream
- Anti-hemorrhoid topical cream drug (Active Comparator): Anti hemorrhoid topical cream as a standard drug 2 cc twice daily for 3 week
  Interventions: Drug: Anti-hemorrhoid topical cream
- Leek topical cream (Active Comparator): Leek (Allium Ampeloprasum Spp.Iranicum) topical cream 2 cc twice daily for 3 weeks
  Interventions: Drug: Leek topical cream

INTERVENTIONS:
Drug: Leek topical cream — Leek (Allium Ampeloprasum Spp.Iranicum) topical cream 2 cc twice daily for 3 weeks
  Other Names: Allium Ampeloprasum Spp.Iranicum topical cream
  Arms: Leek topical cream
Drug: placebo topical cream — placebo topical cream 2 cc twice daily for 3 weeks
  Arms: placebo
Drug: Anti-hemorrhoid topical cream — Anti hemorrhoid topical cream 2 cc twice daily for 3 weeks(This cream consists of lidocaine (5% w/w), hydrocortisone acetate (7.5% w/w), aluminium sub-acetate (3.5% w/w), and zinc oxide (18% w/w). 30 g )
  Arms: Anti-hemorrhoid topical cream drug

SUMMARY:
Purpose of study is evaluation of Allium ampeloprasum Spp.Iranicum cream efficacy in management of symptomatic hemorrhoids in a double blind randomized placebo-control trial

DETAILED DESCRIPTION:
Purpose of study: evaluation of Allium ampeloprasum Spp.Iranicum cream efficacy for the management of hemorrhoids study design:Double blind randomized placebo-control trial, uni-central Study population: Participants having symptomatic hemorrhoids attending Shiraz University of Medical Sciences clinics Inclusion criteria: Patients with symptomatic hemorrhoids(GRADE 1-4) without need to emergency operation according to physical examination Exclusion criteria: Participants having anal fissure or inflammatory bowel disease or history of gastrointestinal cancer Sample size: 75 patients (tree groups) Interventions: Topical Allium ampeloprasum cream/ placebo cream/anti-hemorrhoid cream Time period: 3 week Outcome measures: pain,itching, bleeding, defecate discomfort, total improvement, constipation

ELIGIBILITY:
Inclusion Criteria

* Participants having symptomatic hemorrhoids(GRADE 1-4) without need to emergency operation according to physical examination
* Participants who do not use drugs other than the study drug and the control drug to treat their hemorrhoids during the study period:

Exclusion Criteria:

* Participants having anal fissure or inflammatory bowel disease or history of gastrointestinal cancer
* Participants having hypersensitive predisposition or hypersensitive to Allium ampeloprasum or history of skin hypersensivity
* Female participants under pregnancy or during breastfeeding period
* Participants complicated by serious cardio cerebro vascular diseases, hepatic and renal diseases, diseases of hemopoietic system or neurologic disorders or ascitis g- history of steroid or anticoagulant drug consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
pain (visual analogue scale(0-10)) | 3 weeks
  method of measurement: visual analogue scale(0-10)
bleeding ( questionnaire) | 3 weeks
  method of measurement questionnaire:grade (0-4) that was defined as follow: 0=no symptom, 1= mild, 2=moderate, 3= severe, 4=very severe.
itching ( questionnaire) | 3 weeks
  method of measurement questionnaire: grade (0-4) that was defined as follow: 0=no symptom, 1= mild, 2=moderate, 3= severe, 4=very severe.
defecate discomfort (visual analogue scale(0-10) | 3 weeks
  method of measurement: visual analogue scale(0-10)
total improvement (visual analogue scale(0-10) | 3 weeks
  method of measurement:visual analogue scale(0-10)

SECONDARY OUTCOMES:
constipation (questionnaire) | 3 weeks
  method of measurement: questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ghahramani, Assistant proffessor, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Vice-Chancellery of Research and Technology office, Shiraz University of Medical Sciences, Shiraz, Fars, Iran